## **Protocol Synopsis**

Title: Multicenter Trial of the Sidus Stem-Free Shoulder Arthroplasty System Protocol No.: CIU2012-12E **Sponsor:** Zimmer Inc. **Primary Objectives Objectives:** The primary objectives of this study are to evaluate the safety and efficacy of the Sidus Stem-Free Shoulder System in unilateral primary total shoulder arthroplasty. **Safety** will be evaluated by monitoring the frequency and incidence of device related adverse events or unanticipated adverse device effects (UADEs) in investigational subjects as well as analyzing survivorship using revision or intended revision as an endpoint. Efficacy will be determined by comparing the overall pain and functional performance as well as radiographic investigational subjects with those who received the control devices. The Sidus Stem-Free Shoulder System is indicated for uncemented use Indication/ **Target** in total shoulder arthroplasty, replacing the shoulder joint of subjects **Population:** suffering from severe pain or disability resulting from one or more of the following provided there is adequate bone stock to support the fixation of the implants: Osteoarthritis Posttraumatic arthrosis • Rheumatoid arthritis without humeral metaphyseal defects Previous shoulder surgeries that do not compromise fixation **Study Design:** Multi-center, prospective, historical controlled. **Clinical Phase:** Investigational Device Exemption Protocol / Pre-market 95 subjects will be enrolled in this study at up to 15 centers. Number of **Subjects:** 

## **Protocol Synopsis**

| Title: | Multicenter Trial of the Sidus Stem-Free Shoulder Arthroplasty System |
|---|---|
| Length of Study: | Initial follow-up will be 2 years from the date of enrollment completion to support product approval. Intervals include pre-op, operative, immediate post-op, 6 weeks, 6 months, 1 year, 2 years, and annually until the last subject completes two years of follow-up. |
| Investigational<br>Device System: | <ul> <li>Zimmer Anatomical Shoulder Glenoid</li> <li>Sidus Humeral Head</li> <li>Sidus Stem-Free Anchor</li> </ul> |
| Scores: | <ul> <li>American Shoulder and Elbow Society Standardized Shoulder<br/>Assessment (ASES)</li> <li>SF-12</li> <li>Western Ontario Osteoarthritis Score (WOOS)</li> </ul> |
| Statistical Analysis | |
| Documentation: | Electronic Data Capture. |
| Anticipated<br>Enrollment Date | Zimmer is currently recruiting investigational sites. |

*NOTE:* The investigation described by this protocol involves a significant risk device as defined by the Investigational Device Exemption (IDE) regulation, Part 812, of the Code of Federal Regulations, Food and Drug Administration (FDA).



Sidus Stem-Free Shoulder